CLINICAL TRIAL: NCT01465958
Title: An Open-label, Single-sequence, Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Subcutaneous GAMUNEX®-C in Pediatric Subjects With Primary Immunodeficiency
Brief Title: Pharmacokinetics, Safety, and Tolerability of Subcutaneous GAMUNEX-C in Pediatric Subjects With Primary Immunodeficiency
Acronym: KIDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: T5004-401
Record Dates: First submitted 2011-10-24; First posted 2011-11-07 (Estimated); Results first posted 2015-01-28 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-02

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous GAMUNEX-C (Active Comparator)
  Interventions: Biological: GAMUNEX-C
- Subcutaneous GAMUNEX-C (Experimental)
  Interventions: Biological: GAMUNEX-C

INTERVENTIONS:
Biological: GAMUNEX-C — GAMUNEX-C Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified, Intravenous Administration: 200-600 mg/kg per intravenous infusion every 3-4 weeks
  Arms: Intravenous GAMUNEX-C
Biological: GAMUNEX-C — GAMUNEX-C Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified, Subcutaneous Administration: weekly subcutaneous infusion at a mg/kg dose based on subject's intravenous dose and dosing interval x 1.37 conversion factor
  Arms: Subcutaneous GAMUNEX-C

SUMMARY:
The purpose of this open-label study is to evaluate the pharmacokinetics, safety, and tolerability of subcutaneously (SC; under the skin) administered GAMUNEX-C compared to intravenously (IV; through the vein) administered GAMUNEX-C in subjects 2-16 years of age with Primary Immunodeficiency.

DETAILED DESCRIPTION:
This study was a multi-center, open-label, single-sequence, crossover study to evaluate the pharmacokinetics (PK), safety and tolerability of SC-administered GAMUNEX-C in pediatric PI subjects (ages 2-16). The study consisted of a Screening Phase, Run-in Phase, two treatment phases (an IV Phase and a SC Phase), and an End of Study/Early Termination (EOS/ET) visit. Run-in phase: 3 - 4 months, IV Phase: ~ 4 - 5 weeks, SC Phase: 12 weeks, and End of Study/Early Termination (EOS/ET) visit: one week after SC Week #12.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2-16 years old, inclusive.
* Documented and confirmed pre-existing diagnosis of PI with features of hypogammaglobulinemia requiring immunoglobulin replacement.
* Currently on IgG replacement therapy with a serum IgG trough concentration of ≥ 500 mg/dL at the Screening Visit.
* Adequate normal skin to allow for SC infusions.
* Signs an assent form, if applicable (per Institutional Review Board [IRB] requirements). Parent or legal guardian must sign an informed consent form.
* Females of childbearing potential must have a negative urine pregnancy test result and must practice an effective form of contraception (which may include abstinence).

Exclusion Criteria:

* History of anaphylaxis or severe systemic response to an immunoglobulin or blood product.
* History of blistering skin disease, clinically significant thrombocytopenia, bleeding disorder, recurrent skin infections or other disorders where subcutaneous therapy could be contraindicated.
* Has a specific antibody deficiency disorder, IgG subclass deficiency, or transient hypogammaglobulinemia of infancy.
* History of severe adverse reaction to parenteral products containing immunoglobulin A (IgA).
* Significant proteinuria and/or has a history of acute renal failure and/or severe renal impairment (serum creatinine more than 2.5 times the upper limit of normal [ULN] for age and gender) and/or is on dialysis.
* Known substance or prescription drug abuse in the past 12 months.
* Acquired medical condition that is known to cause secondary immune deficiency.
* Receiving any of the following medications: systemic corticosteroids (long term daily, >1 mg of prednisone equivalent/kg/day for >30 days) (intermittent courses would not exclude subject); immunosuppressants (i.e., antimetabolites and systemic calcineurin inhibitors; NOTE: inhaled steroids are allowed); or immunomodulators.
* Non-controlled arterial hypertension at a level of ≥ the 90th percentile blood pressure (either systolic or diastolic) for age and height (based on http://www.nhlbi.nih.gov/guidelines/hypertension/child_tbl.pdf ).
* History or current diagnosis of thrombotic episodes; venous thrombus that occurred in association with a medical device > 2 years prior to screening are allowed.
* Currently receiving anti-coagulation therapy.
* History of Kawasaki disease.
* Participated in another clinical trial involving exposure to an investigational product or device within 30 days prior to screening (imaging studies without investigative treatments are permitted) or has received any investigational blood product within the previous 3 months.
* Unable or unwilling to comply with any aspect of the protocol, including blood sampling and completion of the Infusion Site Reactions pages in the SC Infusion Diary.
* In the opinion of the Investigator the subject may have compliance problems with the protocol and the procedures of the protocol.
* Pregnant or lactating.
* Clinical evidence of any significant acute or chronic disease that, in the opinion of the Investigator, may interfere with successful completion of the study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Heimall J, Chen J, Church JA, Griffin R, Melamed I, Kleiner GI. Pharmacokinetics, Safety, and Tolerability of Subcutaneous Immune Globulin Injection (Human), 10 % Caprylate/Chromatography Purified (GAMUNEX(R)-C) in Pediatric Patients with Primary Immunodeficiency Disease. J Clin Immunol. 2016 Aug;36(6):600-9. doi: 10.1007/s10875-016-0311-4. Epub 2016 Jun 25. PMID 27342758

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 subjects were screened for participation in this study. After screening, one subject discontinued the study and did not receive study drug. Eleven subjects entered the Run-in phase. One subject entered intravenous Gamunex-C phase directly. A total of 11 subjects entered the IV phase and subsequently entered the SC phase.
Groups:
- Intravenous GAMUNEX-C: GAMUNEX-C: Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified: In the Run-in Phase, subjects received intravenous infusions of Gamunex-C at a dose between 200 to 600 mg/kg every three or four weeks for 3 months. In the subsequent IV phase, subjects received two IV infusions of Gamunex-C at a dose between 200 to 600 mg/kg for four to five weeks.
- Subcutaneous GAMUNEX-C: GAMUNEX-C: Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified: weekly subcutaneous infusion at a mg/kg dose based on intravenous dose of subject and dosing interval x 1.37 conversion factor for 12 weeks.
Period: Run-in Phase
Arm/Group | Intravenous GAMUNEX-C | Subcutaneous GAMUNEX-C
Started | 11 | 0
Completed | 10 | 0
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Intravenous (IV) Phase
Arm/Group | Intravenous GAMUNEX-C | Subcutaneous GAMUNEX-C
Started | 11 (One subject entered the IV phase directly.) | 0
Completed | 11 | 0
Not Completed | 0 | 0
Period: Subcutaneous (SC) Phase
Arm/Group | Intravenous GAMUNEX-C | Subcutaneous GAMUNEX-C
Started | 0 (After completing the intravenous (IV) phase, subjects entered the subcutaneous (SC) phase.) | 11 (Eleven subjects completed the IV phase and entered the SC phase.)
Completed | 0 | 10
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All 12 enrolled subjects who were infused with any amount of study drug (GAMUNEX-C) were included in the safety population. The demographic data of the safety population are provided.
Groups:
- Safety Population: The safety population consisted of all subjects who received any amount of GAMUNEX-C. In the Run-in Phase, subjects received intravenous infusions of Gamunex-C at a dose between 200 to 600 mg/kg every three or four weeks for 3 months. In the subsequent IV phase, subjects received two IV infusions of Gamunex-C at a dose between 200 to 600 mg/kg for four to five weeks. In the SC Phase, subjects received weekly subcutaneous infusion of Gamunex-C at a mg/kg dose based on intravenous dose of the subject and dosing interval x 1.37 conversion factor for 12 weeks.
Arm/Group | Safety Population
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Steady-state Area Under the Curve (AUC) for Serum Total Immunoglobulin (IgG)
Description: Steady-state area under the curve (AUC): For the IV phase, the mean adjusted AUC was calculated for all 11 subjects, which included subjects on both 3 and 4 week intravenous (IV) dosing schedules and who had sufficient immunoglobulin G (IgG) data. For the SC phase, the mean AUC was calculated for 10 subjects on weekly subcutaneous (SC) administration and who had sufficient IgG data.
Time Frame: 4 to 5 weeks for IV administration; 12 weeks for SC administration
Population: The PK population included the subjects with the availability of sufficient pharmacokinetics (PK) data to calculate area under the curve (AUC) for either the IV or SC phases.
Measure: Mean (Full Range); unit: h*mg/dL
Groups:
- Intravenous GAMUNEX-C: GAMUNEX-C: Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified, Intravenous Administration: In the IV phase, subjects received two IV infusions of Gamunex-C at a dose between 200 to 600 mg/kg for four to five weeks.
- Subcutaneous GAMUNEX-C: GAMUNEX-C: Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified, Subcutaneous Administration: weekly subcutaneous infusion at a mg/kg dose based on intravenous dose and dosing interval x 1.37 conversion factor for 12 weeks.
Arm/Group | Intravenous GAMUNEX-C | Subcutaneous GAMUNEX-C
Number analyzed (Participants) | 11 | 10
h*mg/dL | 216873.7 [162277.0 to 291785.0] | 230830.0 [187577.0 to 303913.0]

2. Primary Outcome: Mean Trough of Serum Total IgG
Description: Mean trough serum total IgG values were calculated for each subject for the IV Phase (IV #1 and IV #2) and the SC phase (SC Weeks #9 and #12, and End of Treatment/Early termination visit). Mean trough concentration values of serum total IgG during the IV and SC phases were calculated based on the IgG population (subjects who received any amount of study drug and had serum total IgG concentration data).
Time Frame: 4 - 5 weeks of IV administration and 12 weeks for SC administration
Population: The IgG Population was used to calculate the trough serum concentrations. The IgG population consisted of all subjects who received any amount of GAMUNEX-C and had any serum total IgG concentration data.
Measure: Mean (Full Range); unit: mg/dL
Groups:
- Intravenous GAMUNEX-C: GAMUNEX-C: Immune Globulin Injection (Human), 10%, Caprylate/Chromatography Purified, Intravenous Administration: Two intravenous infusions at a dose of 200-600 mg/kg per intravenous infusion every 3-4 weeks for 4 to 5 weeks.
Arm/Group | Intravenous GAMUNEX-C | Subcutaneous GAMUNEX-C
Number analyzed (Participants) | 11 | 10
mg/dL | 997.2 [784 to 1320] | 1325.0 [1077 to 1690]

ADVERSE EVENTS:
Time Frame: Eligible subjects entered into a 3-month Run-in Phase to receive GAMUNEX-C intravenous infusions. Subjects who completed the Run-in Phase then entered the Intravenous (IV) phase (4 - 5 weeks) followed by the subcutaneous (SC) phase (12 weeks).
Arm/Group | Intravenous GAMUNEX-C | Subcutaneous GAMUNEX-C
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/11
Other Adverse Events (participants affected / at risk) | 10/12 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous GAMUNEX-C (N=12) | Subcutaneous GAMUNEX-C (N=11)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — One subject experienced a serious adverse event (SAE) of lower limb fracture (verbatim term: spiral fracture of right tibia and fibula) during the SC phase that was "not related" to GAMUNEX-C administration.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous GAMUNEX-C (N=12) | Subcutaneous GAMUNEX-C (N=11)
Infusion site erythema (General disorders) | 0 | 7 (11)
infusion site pain (General disorders) | 0 | 6 (9)
Infusion site pruritus (General disorders) | 0 | 6 (19)
Infusion site discomfort (General disorders) | 0 | 3 (12)
Infusion site haematoma (General disorders) | 0 | 3 (10)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Infusion site swelling (General disorders) | 0 | 2 (4)
Pyrexia (Nervous system disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1 (1)
Corona virus infection (Infections and infestations) | 0 | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Gastroenteritis (Infections and infestations) | 0 | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 0 | 1 (1)
Infusion site haemorrhage (General disorders) | 0 | 1 (1)
Infusion site induration (General disorders) | 0 | 1 (2)
Infusion site inflammation (General disorders) | 0 | 1 (1)
Infusion site warmth (General disorders) | 0 | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Skin chapped (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Cellulitis (Infections and infestations) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Croup infectious (Infections and infestations) | 1 (1) | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Fatigue (General disorders) | 1 (1) | 0
Gastrostomy tube insertion (Surgical and medical procedures) | 1 (1) | 0
Incontinence (Renal and urinary disorders) | 1 (1) | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0
Learning disability (Social circumstances) | 1 (1) | 0
Migraine (Nervous system disorders) | 1 (1) | 0
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Seasonal allergy (Immune system disorders) | 1 (1) | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Viral pharyngitis (Infections and infestations) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less